CLINICAL TRIAL: NCT03150667
Title: Pragmatic Randomized Controlled Trial Comparing Treatment Effectiveness of Guideline Indicated Anti-platelet Therapy for Acute Coronary Syndrome in Patients With Chronic Kidney Disease
Brief Title: Study Comparing Treatment Effectiveness of Guideline Indicated APT for ACS in Patients With CKD
Acronym: CPRS-CKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Subhash Banerjee, Chief, Division of Cardiology, North Texas Veterans Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-041
Record Dates: First submitted 2017-05-05; First posted 2017-05-12 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Chronic Kidney Diseases; Acute Coronary Syndrome
MeSH Terms: conditions — Renal Insufficiency, Chronic; Acute Coronary Syndrome | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ticagrelor Arm (Active Comparator): Eligible patients randomized to the Ticagrelor arm will receive open label drug at a dose selected by their providers along with 81mg aspirin. These patients will be followed for 1 year through chart review for events. For event free patients, a phone follow-up will be done at the end of 1 year to record events These events be documented in the medical records.
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator): Eligible patients randomized to the Clopidogrel arm will receive open label drug at a dose selected by their providers along with 81mg aspirin. These patients will be followed for 1 year through chart review for events. For event free patients, a phone follow-up will be done at the end of 1 year to record events These events be documented in the medical records
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — Ticagrelor in patients with CKD presenting with ACS.
  Other Names: Brilinta
  Arms: Ticagrelor Arm
Drug: Clopidogrel — Clopidogrel in patients with CKD presenting with ACS.
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
To compare clinical outcomes in patients with chronic kidney disease (CKD) presenting with an acute coronary syndrome (ACS) treated with clopidogrel or ticagrelor (both FDA approved and guideline indicated drugs for treating these patients upstream managed medically or with coronary revascularization).

DETAILED DESCRIPTION:
The purpose of this trial is to see if ticagrelor is a better antiplatelet treatment option than clopidogrel for dual antiplatelet therapy (with aspirin) in chronic kidney disease (CKD) patients presenting with acute coronary syndrome (ACS). This study will be a comparative effectiveness trial of the two guideline-based treatments for patients with ACS with CKD, who are at a significantly higher risk of mortality and morbidity and often receive sub-optimal treatment. Ticagrelor and clopidogrel are the only two drugs in ACS that are approved for upstream (on admission) use both in CKD and non-CKD patients who are managed both medically (conservatively) or with coronary revascularization (with PCI-percutaneous coronary revascularization or CABG-coronary artery bypass graft surgery). Both of these drugs are not cleared renally and do not require dose adjustments in any stage of CKD.

Moreover, as a significant majority of CKD patients presenting with ACS are initially cared for by internists, hospitalists, and nephrologists, execution of this study at VA hospitals will strengthen collaboration between these specialties with cardiology and help adopt best practice pathways across multiple services participating in the care of this high-risk patient population. Finally, the study and its findings will for the first time provide randomized clinical trial evidence to guide the care of CKD patients with ACS who are at a high risk for both recurrent ischemia and bleeding complications.

Hypothesis to be tested: The Investigators hypothesize that use of guideline-indicated dual antiplatelet therapy (DAPT) with ticagrelor compared to clopidogrel in CKD patients presenting with ACS will reduce ischemic cardiovascular events at 1 year, additionally without a significant increase in severe bleeding (Bleeding Associated Research Consortium or BARC >3 category) over the same period. This hypothesis is based on prior subgroup analysis of published studies.

Randomized patients will be followed for 1 year from date of admission and events recorded through chart review. For patients who are event free, a phone follow-up will be done at the end of 1 year to note events, which will be recorded on the medical chart as well.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission with non-emergent ACS qualifying diagnosis: chest pain, unstable angina or NSTEMI
* A decision to prescribe clopidogrel or ticagrelor in addition to aspirin (DAPT-dual antiplatelet therapy) by the attending physician
* A eGFR< 60 mL/min per 1.73 m.2 (as defined in the EMR or CPRS reported results)

Exclusion Criteria:

* Diagnosis of ST Elevation Myocardial Infarction (STEMI) at admission
* History of intra-cranial hemorrhage
* Bleeding requiring hospitalization, surgery, or transfusion within the past 3 months
* Life expectancy in the opinion of the provider < 6 months
* Chronic antithrombotic therapy
* Known allergy to clopidogrel or ticagrelor
* Patients on hemodialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2020-04-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of all-cause mortality, non-fatal myocardial infarction (MI), or ischemic stroke | 1 year from date of admission
  Occurrence of all-cause mortality, non-fatal myocardial infarction (MI), or ischemic stroke

SECONDARY OUTCOMES:
Occurrence of bleeding | 1 year from date of admission
  Incidence of BARC >3 bleeding over a period of 1-year from hospital admission
Need for ischemia driven urgent coronary revascularization | 1 year from date of admission
  Need for ischemia driven urgent coronary revascularization (UCR) over a period of 1-year from hospital admission
Occurrence of MACE events | 1 year from date of admission
  Comparison of 12-month post-randomization MACE events, a composite of all-cause death, MI, ischemic stroke, or UCR in participant groups
Length of hospital stay and readmission | 1 year from date of admission
  Post-PCI length of hospital stay and readmission ≤ 1 year of initial discharge

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Durham VA Medical Center, Durham, North Carolina
  - VA North Texas Health Care System, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Best PJ, Lennon R, Ting HH, Bell MR, Rihal CS, Holmes DR, Berger PB. The impact of renal insufficiency on clinical outcomes in patients undergoing percutaneous coronary interventions. J Am Coll Cardiol. 2002 Apr 3;39(7):1113-9. doi: 10.1016/s0735-1097(02)01745-x. PMID 11923033
- [Background] Best PJ, Steinhubl SR, Berger PB, Dasgupta A, Brennan DM, Szczech LA, Califf RM, Topol EJ; CREDO Investigators. The efficacy and safety of short- and long-term dual antiplatelet therapy in patients with mild or moderate chronic kidney disease: results from the Clopidogrel for the Reduction of Events During Observation (CREDO) trial. Am Heart J. 2008 Apr;155(4):687-93. doi: 10.1016/j.ahj.2007.10.046. Epub 2008 Feb 21. PMID 18371477
- [Background] Bonello L, De Labriolle A, Roy P, Steinberg DH, Okabe T, Pinto Slottow TL, Xue Z, Torguson R, Suddath WO, Satler LF, Kent KM, Pichard AD, Lindsay J, Waksman R. Impact of optimal medical therapy and revascularization on outcome of patients with chronic kidney disease and on dialysis who presented with acute coronary syndrome. Am J Cardiol. 2008 Sep 1;102(5):535-40. doi: 10.1016/j.amjcard.2008.04.040. Epub 2008 Jun 26. PMID 18721508
- [Background] Charytan D, Kuntz RE. The exclusion of patients with chronic kidney disease from clinical trials in coronary artery disease. Kidney Int. 2006 Dec;70(11):2021-30. doi: 10.1038/sj.ki.5001934. Epub 2006 Oct 18. PMID 17051142
- [Background] Dasgupta A, Steinhubl SR, Bhatt DL, Berger PB, Shao M, Mak KH, Fox KA, Montalescot G, Weber MA, Haffner SM, Dimas AP, Steg PG, Topol EJ; CHARISMA Investigators. Clinical outcomes of patients with diabetic nephropathy randomized to clopidogrel plus aspirin versus aspirin alone (a post hoc analysis of the clopidogrel for high atherothrombotic risk and ischemic stabilization, management, and avoidance [CHARISMA] trial). Am J Cardiol. 2009 May 15;103(10):1359-63. doi: 10.1016/j.amjcard.2009.01.342. Epub 2009 Apr 1. PMID 19427428
- [Background] Fox CS, Muntner P, Chen AY, Alexander KP, Roe MT, Cannon CP, Saucedo JF, Kontos MC, Wiviott SD; Acute Coronary Treatment and Intervention Outcomes Network registry. Use of evidence-based therapies in short-term outcomes of ST-segment elevation myocardial infarction and non-ST-segment elevation myocardial infarction in patients with chronic kidney disease: a report from the National Cardiovascular Data Acute Coronary Treatment and Intervention Outcomes Network registry. Circulation. 2010 Jan 26;121(3):357-65. doi: 10.1161/CIRCULATIONAHA.109.865352. Epub 2010 Jan 11. PMID 20065168
- [Background] Hwang SJ, Lin MY, Chen HC, Hwang SC, Yang WC, Hsu CC, Chiu HC, Mau LW. Increased risk of mortality in the elderly population with late-stage chronic kidney disease: a cohort study in Taiwan. Nephrol Dial Transplant. 2008 Oct;23(10):3192-8. doi: 10.1093/ndt/gfn222. Epub 2008 May 1. PMID 18450830
- [Background] Iakovou I, Schmidt T, Bonizzoni E, Ge L, Sangiorgi GM, Stankovic G, Airoldi F, Chieffo A, Montorfano M, Carlino M, Michev I, Corvaja N, Briguori C, Gerckens U, Grube E, Colombo A. Incidence, predictors, and outcome of thrombosis after successful implantation of drug-eluting stents. JAMA. 2005 May 4;293(17):2126-30. doi: 10.1001/jama.293.17.2126. PMID 15870416
- [Background] James MT, Pannu N. Early-invasive strategies for the management of coronary heart disease in chronic kidney disease: is acute kidney injury a consideration? Curr Opin Nephrol Hypertens. 2014 May;23(3):283-90. doi: 10.1097/01.mnh.0000444819.03121.4b. PMID 24662983
- [Derived] Natale P, Palmer SC, Saglimbene VM, Ruospo M, Razavian M, Craig JC, Jardine MJ, Webster AC, Strippoli GF. Antiplatelet agents for chronic kidney disease. Cochrane Database Syst Rev. 2022 Feb 28;2(2):CD008834. doi: 10.1002/14651858.CD008834.pub4. PMID 35224730